CLINICAL TRIAL: NCT05237193
Title: A Prospective, Multi-centre, Single-blinded Study of UCAD for Diagnosing Benign or Malignant Biliary Obstruction and Follow-up
Brief Title: A Prospective Study of UCAD for Diagnosing Benign or Malignant Biliary Obstruction and Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); Changhai Hospital (Other); Shanghai Changzheng Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Jiangsu Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Zhejiang University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Hospital of Jilin University (Other); West China Hospital (Other); Southwest Hospital, China (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: XH-22-001
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-05

CONDITIONS: Biliary Tract Neoplasms; Pancreatic Carcinoma; Gallbladder Cancer; Pancreatic Head Carcinoma
Keywords: diagnosis; follow-up
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms; Gallbladder Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from bile tract exfoliated cells will be analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- malignant biliary obstruction: Pre-surgery patients with malignant biliary obstruction will be the experimental group to determine the sensitivity and specificity of UCAD analysis, the result will be compared with cytology.
  Interventions: Diagnostic Test: The level of CIN
- Benign biliary obstruction: Patients being treated for other biliary diseases but without any tumor will provide a negative control to provide data for determining the sensitivity and specificity of UCAD analysis.
  Interventions: Diagnostic Test: The level of CIN

INTERVENTIONS:
Diagnostic Test: The level of CIN — The extracted DNA from bile will be analyzed by UCAD to determine the level of CIN. And the patient will be followed for up to 2 years.

SUMMARY:
Chromosomal instability (CIN) refers to ongoing chromosome segregation errors throughout consecutive cell divisions. CIN is a hallmark of human cancer, and it is associated with poor prognosis, metastasis, and therapeutic resistance. Analyzing CIN of the DNA extracted from bile tract exfoliated cells in bile samples seems a promising method for diagnosing, monitoring, and predicting the prognosis of patients with malignant biliary obstruction, including biliary tract cancer (BTC), pancreatic head carcinoma. CIN can be assessed using experimental techniques such as bulk DNA sequencing, fluorescence in situ hybridization (FISH), or conventional karyotyping. However, these techniques are either time-consuming or non-specific. The investigators here intend to study whether a new method named Ultrasensitive Chromosomal Aneuploidy Detection (UCAD), which is based on low-coverage whole-genome sequencing, can be used to analyze CIN thus helping diagnose malignant biliary obstruction and assessing follow-up.

DETAILED DESCRIPTION:
CIN results from errors in chromosome segregation during mitosis, leading to structural and numerical chromosomal abnormalities. It will generate genomic heterogeneity that acts as a substrate for natural selection. Furthermore, it is proved that tumors with aneuploidies and polyploidy resulting from whole-genome doubling are related to metastasis, treatment resistance, and decreased overall survival. It is estimated that 60%-80% of human tumors exhibit chromosomal abnormalities suggestive of CIN. CIN positively correlates with tumor stage and is enriched in relapsed as well as metastatic tumor specimens. Due to the ubiquity of CIN in cancer cells, it is a potentially non-invasive way to detect CIN in the bile tract exfoliated cells in bile samples for diagnosing and monitoring malignant biliary obstruction patients. UCAD is a new method to detect CIN in the DNA sample from patients, including extracting DNA from bile, analyzing DNA by low-coverage whole-genome sequencing, processing the data by bio-information techniques, and finally optimizing the management of malignant biliary obstruction patients. The investigators intended to conduct a prospective, single-blinded study by analyzing bile samples from malignant biliary obstruction patients and control groups without any tumor in the biliary system or other organs to compare the specificity and sensitivity of the UCAD test for diagnosing malignant biliary obstruction to other modalities, such as bile cytology. The investigators also intend to investigate the potential of UCAD in malignant biliary obstruction patient follow-up by analyzing the CIN level and following malignant biliary obstruction patients for up to 2 years to determine if there is a correlation between CIN level and patient prognosis

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with malignant biliary obstruction and planned to undergo ERCP(endoscopic retrograde cholangiopancreatography), PTCS(percutaneous transhepatic cholangioscopy) or surgery.
* Malignant biliary obstruction patients confirmed by operation or biopsy.
* Participants without any tumor disease and willing to attend the study.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Patients diagnosed with malignant biliary obstruction and planned to undergo ERCP, PTCS or surgery.
* Malignant biliary obstruction patients confirmed by operation or biopsy.
* Participants without any tumor disease and willing to attend the study.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with malignant biliary obstruction or participants in control group from February 2022 till the end of this study in 11 hospitals including Xinhua Hospital, Shanghai Zhongshan Hospital, Ruijin Hospital, Changhai Hospital, Shanghai Changzheng Hospital, Eastern Hepatobiliary Surgery Hospital, The First Affiliated Hospital of Xi'an Jiaotong University, Jiangsu Provincial Hospital, The Third Affiliated Hospital of Sun Yat-Sen University, Tianjin Medical University Second Hospital, First Affiliated Hospital of Zhejiang University.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of UCAD analysis | through study completion, an average of 30 months
  number of patients "declared positive" with the UCAD test among the patients who suffered from malignant biliary obstruction and number of patients "declared negative" with the UCAD test among the patients without cancer
Assess the value of UCAD for malignant biliary obstruction patient follow-up | through study completion, an average of 30 months
  Compare the CIN level with the patient information gathered by follow-up to determine whether there is a correlation between CIN level and patient prognosis , like PFS(progression-free survival), five-year survival rate.

SECONDARY OUTCOMES:
Identification of the correlation between the level of CIN and the grade of the tumor sample | through study completion, an average of 30 months
  level of CIN in the bile sample compared with the grade of the tumor confirmed by histopathologic examination, like Grade 1-4.
Identification of the correlation between the level of CIN and the stage of the tumor sample | through study completion, an average of 30 months
  level of CIN in the bile sample compared with the TNM stage of the tumor confirmed by histopathologic examination, like Stage 0-IV.
Comparison of the sensitivity and specificity of the UCAD analysis versus bile cytology | through study completion, an average of 30 months
  number of patients "declared positive" with the UCAD analysis versus patients "declared positive" with the bile cytology and number of patients "declared negative" with the UCAD analysis versus patients " declared negative " with the bile cytology

CONTACTS AND LOCATIONS:
Overall Officials: Jiandong Jiandong, M.D., Ph.D., Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will try to protect the information of the included participants

REFERENCES:
- [Background] Hieronymus H, Murali R, Tin A, Yadav K, Abida W, Moller H, Berney D, Scher H, Carver B, Scardino P, Schultz N, Taylor B, Vickers A, Cuzick J, Sawyers CL. Tumor copy number alteration burden is a pan-cancer prognostic factor associated with recurrence and death. Elife. 2018 Sep 4;7:e37294. doi: 10.7554/eLife.37294. PMID 30178746
- [Background] Bakhoum SF, Ngo B, Laughney AM, Cavallo JA, Murphy CJ, Ly P, Shah P, Sriram RK, Watkins TBK, Taunk NK, Duran M, Pauli C, Shaw C, Chadalavada K, Rajasekhar VK, Genovese G, Venkatesan S, Birkbak NJ, McGranahan N, Lundquist M, LaPlant Q, Healey JH, Elemento O, Chung CH, Lee NY, Imielenski M, Nanjangud G, Pe'er D, Cleveland DW, Powell SN, Lammerding J, Swanton C, Cantley LC. Chromosomal instability drives metastasis through a cytosolic DNA response. Nature. 2018 Jan 25;553(7689):467-472. doi: 10.1038/nature25432. Epub 2018 Jan 17. PMID 29342134